CLINICAL TRIAL: NCT03197792
Title: Perioperative Transesophageal Portal Vein Pulsatility as a Predictor of Persistent Organ Dysfunction Plus Death 7 Days After Pulmonary Endarterectomy
Brief Title: Perioperative Portal Vein Pulsatility as a Postoperative Prognostic Indicator in Pulmonary Endarterectomy
Acronym: PVP-ETO-CPC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Chirurgical Marie Lannelongue (Other)
Responsible Party: Principal Investigator, Olaf Mercier, MD, PhD, Professor of thoracic surgery, Centre Chirurgical Marie Lannelongue
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: P17-37813005
Record Dates: First submitted 2017-05-21; First posted 2017-06-23 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Pulmonary Hypertension; Thromboembolism, Pulmonary; Perioperative/Postoperative Complications; Venous Hypertension; Cardiac Failure
Keywords: Transesophageal ultrasound; TEE; Portal vein pulsatility; Splenic vein pulsatility; Venous congestion; Strain; Right ventricular dysfunction; Pulmonary hypertension; Venous hypertension
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Embolism; Postoperative Complications; Heart Failure; Hyperemia; Sprains and Strains; Ventricular Dysfunction, Right

STUDY DESIGN:
Intervention Model Description: Patients with chronic post-embolic pulmonary hypertension eligible to pulmonary endarterectomy surgery will be evaluated for venous congestion and right ventricular failure after weaning of cardiopulmonary bypass, and followed until the 7th postoperative day for the development of postoperative organ dysfunction and/or death.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pulmonary endarterectomy patients (Experimental): All patients
  Interventions: Other: All patients

INTERVENTIONS:
Other: All patients — TEE is performed before cardiopulmonary bypass (before the opening of the pericardium, if possible) and immediately after weaning from cardiopulmonary bypass and optimization of the hemodynamic status by the attending anesthesiologist. A detailed ultrasound examination including portal vein pulsatility, splenic vein pulsatility, right and left ventricular global longitudinal strain and right and left systolic and diastolic function is recorded. A measure of portal vein pulsatility using TTE is also recorded before the onset of general anesthesia and on the morning of the 7th postoperative day.
  On the 7th postoperative day, the investigators will evaluate for the presence of the primary outcome, POD + death.

SUMMARY:
The investigators aim to evaluate the utility of portal vein pulsatility as a predictor of the composite outcome of persistent organ dysfunction plus death in patients undergoing elective or urgent pulmonary endarterectomy for thromboembolic pulmonary hypertension. The investigators' hypothesis is that the portal vein pulsatility fraction, measured using transesophageal echocardiography immediately after weaning of cardiopulmonary bypass, is proportional to the risk of developing subsequent end-organ dysfunction in the postoperative setting.

DETAILED DESCRIPTION:
While transesophageal echocardiography is recommended in patients with known or suspected cardiovascular pathology which may impact outcomes, no study has evaluated it's perioperative use in pulmonary endarterectomy surgery.

Most pulmonary endarterectomy patients suffer from severe pulmonary hypertension, right heart dysfunction and central venous hypertension. Postoperative complications are closely related to the importance of residual postoperative pulmonary hypertension and right ventricular dysfunction. A portal vein pulsatility fraction of 50% or more in the perioperative setting might indicate right ventricular dysfunction and/or hypervolemia-related severe venous congestion, which may be responsible for multiple organ dysfunction and significant morbidity or mortality in critically ill patients.

The investigators believe pulmonary endarterectomy patients with a high portal vein pulsatility fraction immediately after weaning from cardiopulmonary bypass have a greater risk of developing postoperative persistent organ dysfunction and/or death. In this prospective descriptive study, the investigators will evaluate portal vein pulsatility as a predictor of the composite outcome of persistent organ dysfunction plus death 7 days after pulmonary endarterectomy.

Left and right global longitudinal strain after weaning from cardiopulmonary bypass will also be evaluated as potential indicators of a higher risk of persistent organ dysfunction plus death 7 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Elective or urgent pulmonary endarterectomy

Exclusion Criteria:

* absolute or relative contraindication to the use of transesophageal echocardiography,
* hepatic cirrhosis,
* portal vein thrombosis,
* concomitant coronary artery bypass grafting,
* patient refusal or unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2017-05-26 (Actual); Primary Completion 2018-05-24 (Actual); Study Completion 2019-05-24 (Estimated)

PRIMARY OUTCOMES:
Persistent organ dysfunction plus death (POD + death) 7 days after surgery | On the morning of the 7th postoperative day
  POD + death, defined as death or one of the following criterias (yes or no) present on the 7th postoperative day : (1) mechanical ventilation (excluding non-invasive ventilation) without breaks for more than 48 hours, (2) ongoing need for vasopressor therapy more than 2 hours per day (dopamine more than 5 mcg/kg/min, phenylephrine more than 50 mcg/min, norepinephrine, epinephrine, vasopressin), (3) ongoing need for mechanical circulatory support such as ECMO or IABP, and (4) continuous renal replacement therapy or new intermittent hemodialysis.

CONTACTS AND LOCATIONS:
Overall Officials: MOORE ALEX, Dr, Principal Investigator — HOPITAL MARIE LANNELONGUE
Locations (1):
- Hopital Marie Lannelongue, Le Plessis-Robinson, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hahn RT, Abraham T, Adams MS, Bruce CJ, Glas KE, Lang RM, Reeves ST, Shanewise JS, Siu SC, Stewart W, Picard MH; American Society of Echocardiography; Society of Cardiovascular Anesthesiologists. Guidelines for performing a comprehensive transesophageal echocardiographic examination: recommendations from the American Society of Echocardiography and the Society of Cardiovascular Anesthesiologists. Anesth Analg. 2014 Jan;118(1):21-68. doi: 10.1213/ANE.0000000000000016. No abstract available. PMID 24356157
- [Background] Jenkins D. Pulmonary endarterectomy: the potentially curative treatment for patients with chronic thromboembolic pulmonary hypertension. Eur Respir Rev. 2015 Jun;24(136):263-71. doi: 10.1183/16000617.00000815. PMID 26028638
- [Background] Dittrich HC, Chow LC, Nicod PH. Early improvement in left ventricular diastolic function after relief of chronic right ventricular pressure overload. Circulation. 1989 Oct;80(4):823-30. doi: 10.1161/01.cir.80.4.823. PMID 2791245
- [Background] Olson N, Brown JP, Kahn AM, Auger WR, Madani MM, Waltman TJ, Blanchard DG. Left ventricular strain and strain rate by 2D speckle tracking in chronic thromboembolic pulmonary hypertension before and after pulmonary thromboendarterectomy. Cardiovasc Ultrasound. 2010 Sep 27;8:43. doi: 10.1186/1476-7120-8-43. PMID 20875129
- [Background] Marston N, Brown JP, Olson N, Auger WR, Madani MM, Wong D, Raisinghani AB, DeMaria AN, Blanchard DG. Right ventricular strain before and after pulmonary thromboendarterectomy in patients with chronic thromboembolic pulmonary hypertension. Echocardiography. 2015 Jul;32(7):1115-21. doi: 10.1111/echo.12812. Epub 2014 Oct 18. PMID 25327878